CLINICAL TRIAL: NCT03835624
Title: Interleukin 33 in Juvenile Idiopathic Arthritis Patients :Relation to Disease State and Muscloskeletal Ultrasound Findings
Brief Title: Interleukin 33 in Juvenile Idiopathic Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Waleed Ahmed Salaheldeen Hassan, Assistant professor, Benha University
Other Study IDs: Benha University
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile Idiopathic Arthritis; Interleukin 33
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples from Juvenile idiopathic arthritis patients and healthy controls and synovial fluid samples from Juvenile idiopathic arthritis patients

GROUPS / COHORTS (2):
- juvenile idiopathic arthritis: about 60 cases of children with juvenile idiopathic arthritis diagnosed according to ILAR classification criteria of juvenile idiopathic arthritis will be recruited from pediatric rheumatology clinic of Benha university hospital serum interleukin 33 and its relative expression in peripheral blood mononuclear cells (PBMNCs) will be measured in their blood samples also IL-33 will be measured in synovial fluid samples
  Interventions: Diagnostic Test: interleukin 33
- control group: about 60 apparently healthy children with comparable age and sex to the patients.
  serum interleukin 33 and its relative expression in PBMNCs will be measured in their bloodsamples.
  Interventions: Diagnostic Test: interleukin 33

INTERVENTIONS:
Diagnostic Test: interleukin 33 — serum and synovial fluid samples will be obtained from patients and serum samples from controls to measure interleukin 33 and its relative mRNA expression in peripheral blood mononuclear cells by PCR
  Other Names: IL-33

SUMMARY:
The aim of this study is to measure serum and synovial fluid levels of IL 33 and its relative mRNA expression in peripheral blood mononuclear cells in juvenile idiopathic arthritis (JIA) patients and to correlate it with the clinical and laboratory characteristics, disease activity and musculoskeletal ultrasound findings.

DETAILED DESCRIPTION:
SUBJECTS AND METHODS

Subjects:This study will be a case-control study including sixty children with juvenile idiopathic arthritis attending pediatric rheumatology clinic of Benha University Hospital and Benha children hospital and thirty apparently healthy children as controls. They will be classified into:

* Group (I) study group:60 cases of children with juvenile idiopathic arthritis.
* Group (II) Control group:60 of apparently healthy children matched for age and sex

A)Full history taking

B) Full clinical examination

C) Clinical assessment of disease activity

D) Laboratory Investigations:

All subjects will be investigated by

1. complete blood count.
2. Erythrocyte sedmentation rate.
3. C-reactive protein .
4. Liver enzymes: ALT and AST.
5. Rheumatoid factor.
6. Antinuclear antibody (ANA).
7. serum ferritin
8. serum and synovial fluid Interleukin 33 by ELISA and its relative expression in peripheral blood mononuclear cells by PCR

E) Musculoskeletal Ultrasound examination

ELIGIBILITY:
Inclusion Criteria:

* Children less than 16 years old diagnosed according to ILAR classification criteria of juvenile idiopathic arthritis

Exclusion Criteria:

* 1-Exclusion other causes of arthritis in children as:

  1. Other autoimmune diseases Vasculitis- SLE- Rheumatic fever- Dermatomyositis- Polymyositis- Enteropathic arthritis- Behcet disease- Sjogren-Scleroderma- Mixed connective diseases
  2. Infectious disease or septic arthritis.
  3. Metabolic diseases.
  4. Endocrine diseases.
  5. Neuropathic diseases.
  6. Heritable bone disease.
  7. Neoplastic diseases including leukemia.
  8. Sarcoidosis.
  9. Familial Mediterranean fever. 2-Exclusion of children with diseases that affect serum level of IL 33 as:

  <!-- -->

  1. Inflammatory diseases of airway e.g asthma
  2. Inflammatory bowel disease
  3. Systemic lupus erythmatosus
  4. Inflammatory skin disease e.g :atopic dermatitis
  5. Cancer

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will be a case-control study including sixty children with juvenile idiopathic arthritis attending pediatric rheumatology clinic of Benha University Hospital and and 60 apparently healthy children as controls.
  They will be classified into:
  * Group (I) study group:60 cases of children with juvenile idiopathic arthritis.
  * Group (II) Control group:60 of apparently healthy children matched for age and sex.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
27 active joints count | through study completion, an average of 4 months
  active arthritis, defined as joint swelling or limitation of movement accompanied by pain and tenderness, assessed in 27 joints
physician's global assessment of disease activity scale | through study completion, an average of 4 months.
  physician's global assessment of disease activity on a 0- 10 cm visual analogue scale (VAS). Higher value indicates worse outcome
parent/patient global assessment of well-being scale | through study completion, an average of 4 months.isit to measure IL33
  parent/patient global assessment of well-being on a 0-10 cm visual analogue scale .Higher value indicates worse outcome
Erythrocyte sedimentation rate (ESR) | through study completion, an average of 4 months
  ESR measured in mm/1st hour by westergren method
The 27-joint Juvenile Arthritis Disease Activity Score (JADAS-27) | through study completion, an average of 4 months
  The JADAS-27 (range 0-57) was computed by summing the scores of four core-set criteria [3]: physician's global assessment of disease activity (PGA) on a 10 cm visual analogue scale (VAS); parent/patient global assessment of well-being on a 10 cm VAS [7]; active arthritis, defined as joint swelling or limitation of movement accompanied by pain and tenderness, assessed in 27 joints; and ESR (mm/h) normalized to a 0-10 scale, using the formula ESR - 20/10, whereby, before the calculation, ESR values <20 mm/h were converted to 0 and ESR values >120 mm/h were converted to 120. A higher JADAS-27 indicates higher disease activity and a lower JADAS-27 indicates lower disease activity
C reactive protein (CRP) | through study completion, an average of 4 months
  CRP measured in mg/L using nephlometry
Serum ferritin level | through study completion, an average of 4 months
  Serum ferritin level measured in ng/mL using elisa
grey scale 10 joint score | through study completion, an average of 4 months
  grey scale musculoskeletal ultrasound including 10-joints (bilateral knee, ankle, wrist, elbow and the 2nd metacarpophalangeal (MCP) joints)
power Doppler 10 joint score | through study completion, an average of 4 months
  power Doppler musculoskeletal ultrasound including 10-joints (bilateral knee, ankle, wrist, elbow and the 2nd metacarpophalangeal (MCP) joints)
rheumatoid factor | through study completion, an average of 4 months
  rheumatoid factor measured in U/ml using latex agglutination test
disease activity for systemic arthritis with active systemic features (and without active arthritis) | through study completion, an average of 4 months
  DISEASE ACTIVITY LEVELS (2 levels) Active fever AND physician global assessment of overall disease activity 7 of 10 Active fever AND systemic features of high disease activity (e.g., significant serositis) that result in physician global assessment of overall disease activity 7 of 10
The Juvenile Arthritis Multidimensional Assessment Report | through study completion, an average of 4 months
  The JAMAR is a questionnaire includes the following 15 sections:
  Assessment of physical function (PF) using 15-items with score 0-45. Higher scores indicating higher degree of disability 2. 21-numbered circle Visual Analogue Scale (VAS) for pain 3. Assessment of the presence of joint pain or swelling.4.Assessment of morning stiffness 5. extra-articular symptoms (fever and rash) 6.disease activity on a 21-circle VAS. 7.disease status. 8. course. 9.medications . 10. side effects. 11.difficulties with medication 12. school/university/work problems. 13. HRQoL 14.patient's overall well-being on a 21-numbered circle VAS. 15. satisfaction with outcome.
disease activity for systemic arthritis with active arthritis (and without active systemic features) | through study completion, an average of 4 months
  Low disease activity (must satisfy all) 4 or fewer active joints, ESR or CRP level normal PGA of disease activity less than4 of, 10 PAGA of well-being 2 of 10 Moderate disease activity (does not satisfy criteria for low or high disease activity) High disease activity (must satisfy at least 3) 8 or more active joints,ESR or CRP level greater than twice upper limit of normal, PGA of disease activity 7 of 10, PAGA of well-being 5 of 10

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Hassan, MD, Principal Investigator — Benha university- Qaluibya- Egypt
Locations (1):
- Benha University Hospital, Banhā, Qalyubia Governorate, Egypt